CLINICAL TRIAL: NCT01489280
Title: Temple Touch Pro (TTP) Non Invasive Continuous Temperature Measurement System.
Acronym: TTP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medisim Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 26-115-630
Record Dates: First submitted 2011-12-07; First posted 2011-12-09 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Body Temperature During Surgery
Keywords: Temple Touch Pro; Medisim; temperature; surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, the body temperatures of men and women undergoing elective surgery will be measured using the Temple Touch Pro. In the operating room, each patient's temperature will be measured with both the Temple Touch Pro and another one or two of the continuous reference methods used clinically for measuring the core temperature.

The Medisim Temple Touch Pro thermometer combines a noninvasive, biocompatible patch and a receiving unit. The former is attached to the skin, while the latter is placed near the patient or the vital signs monitor and receives data from the patch. The core temperature equivalent is displayed. The Medisim Temple Touch Pro is based on the measurements made by conductive sensors that perform skin temperature measurements and then applies a special algorithm in order to calculate the body's temperature.

ELIGIBILITY:
Inclusion Criteria:

The patients will be chosen for the trial if the following criteria are met:

* Male and female patients scheduled to undergo cardiothoracic surgery and major (surgeries scheduled to last more than 90 minutes) abdominal, vascular and general surgery.
* The surgical procedure requires temperature monitoring.
* Informed consent signed by the patient or his legal guardian.

Exclusion Criteria:

The patients will be excluded from the trial if one of the following occurs:

* The medical staff decides that the patient should not participate.
* Unavailable measurement site in case of operations performed in the head area.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ages 0 and up, patients subjected to elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Rambam medical center, Haifa
  - Wolfson Medical Center, Holon